CLINICAL TRIAL: NCT00457496
Title: Effectiveness of a Cognitive and Physical Program in Reducing Headache, Neck and Shoulder Pain: a Workplace Controlled Trial
Brief Title: Effectiveness of a Cognitive and Physical Intervention to Reduce Head and Muscle Pain in Working Communities
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: Compagnia di San Paolo (Other); Turin, Italy (Other); Centro di Riferimento per l'Epidemiologia e la Prev. Oncologica Piemonte (Other); Regione Piemonte (Other)
Responsible Party: Franco Mongini/ Professor and Chairman, Unit of Headache and Facial Pain, Dept. of Clinical Pathophysiology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5147SD2003.0271
Record Dates: First submitted 2007-04-05; First posted 2007-04-06 (Estimated); Last update posted 2008-07-14 (Estimated); Status verified 2008-07

CONDITIONS: Headache Disorders; Headache; Neck Pain; Shoulder Pain
Keywords: Behavior Therapy; Relaxation Techniques; Cognitive Therapy; Exercise Movement Techniques
MeSH Terms: conditions — Headache Disorders; Headache; Neck Pain; Shoulder Pain | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Active Comparator)
  Interventions: Behavioral: Cognitive, behavioral, exercise

INTERVENTIONS:
Behavioral: Cognitive, behavioral, exercise — Relaxation exercises once a day, visual feedback, exercises for neck and shoulder

SUMMARY:
The primary purpose of this study is to evaluate the effectiveness of a workplace cognitive and physical program (Intervention), in reducing the frequency of head and neck pain

DETAILED DESCRIPTION:
Many studies have been performed to assess the efficacy of non invasive physical interventions in the treatment of different types of headache and cervical pain. However the evidence on their effectiveness is still limited and the results of recent studies are conflicting.

The primary objective of this study is to evaluate the effectiveness of a workplace cognitive and physical programme (Intervention) in reducing the frequency of pain involving the head and neck area. The Intervention consists of brief shoulder and neck exercises to be performed several times a day, a relaxation exercise and instructions of how to reduce parafunction and hyperfunction of the craniofacial and cervical muscles during the day.

Comparison(s): Group of employees that will receive a cognitive/physical programme (Intervention), compared to a similar group of employees that will not receive the Intervention (Controls); (frequency of headache and neck and shoulder pain).

ELIGIBILITY:
Inclusion Criteria:

* Subjects employed at the Municipality of Turin ( Registry-Tax office) from the 1th January 2005 that will give informed consent before starting the study.

Exclusion Criteria:

- Because of the pragmatic design, no exclusion criteria are required for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2005-03; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Frequency of headache and neck and shoulder pain after 6 months (monthly frequency, responder rate) | 6 months

SECONDARY OUTCOMES:
Analgesic drug consumption after 6 and 12 months | 12 months
Headache index after 6 and 12 months | 12 months
Neck and shoulder pain index after 6 and 12 months | 12 months
Muscle tenderness at palpation after 6 and 12 months | 12 months
Psychiatric comorbidity and psychosomatic symptoms prevalence | 12 months
Frequency of pain in head/neck area after 12 months in both groups | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Franco Mongini, Professor, Study Chair — University of Turin, Italy; Eugenia Rota, MD, Principal Investigator — University of Turin, Italy; Alessandro Ugolini, DDS, Principal Investigator — University of Turin, Italy; Luca Ferrero, DDS, Principal Investigator — University of Turin, Italy